CLINICAL TRIAL: NCT02048475
Title: Electroencephalogram During Increasing and Decreasing Desflurane Concentration
Brief Title: Electroencephalogram During Desflurane Anaesthesia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: administrative reasons.
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Arvi Yli-Hankala, Professor, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Kotoe _ 2; 2009-014620-36 (EudraCT Number)
Record Dates: First submitted 2013-10-08; First posted 2014-01-29 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Anesthesia
Keywords: desflurane; electroencephalogram
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- desflurane (No Intervention): inhalation concentration
  Interventions: Other: desflurane

INTERVENTIONS:
Other: desflurane — changing concentration

SUMMARY:
To study the behavior of EEG during changing desflurane concentrations.

DETAILED DESCRIPTION:
The concentration of desflurane will be increased to burst suppression EEG level, and thereafter decreased.

ELIGIBILITY:
Inclusion Criteria:

* adult patients

Exclusion Criteria:

* pediatric patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The behavior of EEG indices numbers during the course of anesthesia, with comparison to raw EEG traces | participants will be followed for the duration of surgical anesthesia, an expected average of 1 hour
  How do the EEG indices reflect the clinical evaluation of anesthetic state and the visual appearance of EEG

CONTACTS AND LOCATIONS:
Overall Officials: Arvi M Yli-Hankala, MD, Principal Investigator — Tampere University Hospital